CLINICAL TRIAL: NCT01762943
Title: Neurophysiology of Postpartum Depression in an Experimental Model of Pregnancy and Parturition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other); North Carolina Translational and Clinical Sciences Institute (Other); National Institutes of Health (NIH) (NIH); National Alliance for Research on Schizophrenia and Depression (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-1758; 5R21MH101409 (NIH)
Record Dates: First submitted 2012-11-13; First posted 2013-01-08 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-02

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Leuprolide; Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Women with Postpartum Depression (PPD) (Experimental): 4 monthly (intramuscular) IM injections of leuprolide acetate (Lupron) 3.75 mg; micronized estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day; progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day. Participants will also receive placebo.
  Interventions: Drug: Leuprolide Acetate; Drug: Micronized estradiol; Drug: Progesterone
- Women without any psychiatric history (Control) (Experimental): 4 monthly (intramuscular) IM injections of leuprolide acetate (Lupron) 3.75 mg; micronized estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day; progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day. Participants will also receive placebo.
  Interventions: Drug: Leuprolide Acetate; Drug: Micronized estradiol; Drug: Progesterone

INTERVENTIONS:
Drug: Leuprolide Acetate — All subjects will receive one IM injection (3.75 mg) each month for four months.
  Other Names: Lupron
Drug: Micronized estradiol — All participants will receive micronized estradiol daily for eight weeks. Estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day.
  Other Names: Estrace
Drug: Progesterone — All subjects will receive micronized progesterone daily for eight weeks. Progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day.
  Other Names: Micronized progesterone

SUMMARY:
Understanding the neural and biological mechanisms by which reproductive hormones influence mood is critically important for public health given that postpartum depression (PPD) is the leading cause of morbidity and mortality associated with childbirth and has negative effects on infants. Using a hormone-withdrawal challenge to precipitate mood symptoms will improve our ability to identify the biological mechanisms underlying both the triggering of and susceptibility to depressive disorders in women; and will permit the prediction of those at risk for PPD and other reproductive-related mood disorders.

DETAILED DESCRIPTION:
Affective disorders, such as PPD and other reproductive-related mood disorders, are common and constitute a significant burden for women, children, and society. However, little is known about the neurobiological mechanisms underlying depressive disorders in women. The long-term goal of this research is to 1) advance our understanding of the biological mechanisms underlying both the triggering of and susceptibility to depressive disorders in women; and 2) permit the prediction of those at risk for PPD. The objective of the current project is to examine whether those with a past episode of PPD (at "high risk" for recurrence) show differences in emotional arousal and reward processing domains relative to healthy control women (without a history of PPD) under baseline and hormone withdrawal-precipitated conditions. The central hypothesis is that reproductive hormone changes are associated with dysregulation of the neural circuits underlying emotional arousal and reward processing and consequent depressive symptoms in high-risk women. The rationale for the proposed study is that employing a scaled down model of puerperal hormonal events in high-risk women permits the identification of a group of individuals homogeneous for reproductive related affective dysfunction and, hence, the best opportunity for disentangling the specific changes in brain function due to reproductive hormones from those accompanying reproductive hormone-precipitated affective dysfunction. Moreover, identifying a neurophysiologic biomarker for hormone-related affective dysfunction provides a clear pathway for examining mechanisms of susceptibility to affective dysfunction across disorders. The investigators plan to accomplish the objectives of this application by pursuing the following specific aims: 1) to assess the effects of simulated postpartum reproductive hormone withdrawal, compared to baseline, on corticolimbic circuit activation in high-risk and control women; and 2) to examine the effects of reproductive hormone withdrawal, compared to baseline, on reward circuit activation in high-risk and control women. An additional exploratory aim is to identify a neural biomarker, characterized by corticolimbic and reward circuit dysfunction, that can be used to predict the onset of PPD. The proposed study involves experimentally manipulating reproductive hormones in euthymic women to create a scaled down version of the changes that occur at the puerperium. This endocrine manipulation paradigm will be used to examine the neurocircuitry underlying the regulation of affect and reward processing under baseline and hormone withdrawal-precipitated conditions among women who are expected to experience hormone-related affective dysregulation (n=15) and controls (n=15). In short, the investigators expect that relative to baseline, high-risk women will show greater dysregulation in neural circuits responsible for emotion processing and reward processing during hormone withdrawal than low-risk control women. The expected outcome of this research is the identification of neural circuits underlying both the susceptibility to and mediation of hormone-related affective dysfunction. Understanding these neurobiological mechanisms will subsequently improve the ability to identify those at risk for PPD, which may strengthen prevention efforts and ultimately prevent the deleterious effects of maternal depression on offspring.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Women with a history of PPD

1. A history of a major depression episode that occurred within two months of childbirth (as determined by a SCID interview) and remitted at least one year prior to enrollment in the study;
2. has been well for a minimum of one year;
3. a regular menstrual cycle for at least three months;
4. age 22-50;
5. not pregnant, not lactating and in good medical health;
6. medication free (not including birth control pills; participants may opt to temporarily discontinue birth control pills to participate);
7. no history of puerperal suicide attempts or psychotic episodes requiring hospitalization.

Group 2: Healthy Controls

1) Controls will meet all inclusion criteria specified above except they must not have any past or present Axis I diagnosis or evidence of menstrually related mood disorders.

A structured clinical interview (SCID) will be administered to all women prior to study entry. Any woman with a current axis I psychiatric diagnosis will be excluded from participating in this protocol.

Exclusion Criteria:

Patients will not be permitted to enter this protocol if they have important clinical or laboratory abnormalities including any of the following:

* current axis I psychiatric diagnosis
* endometriosis;
* undiagnosed enlargement of the ovaries;
* liver disease;
* breast cancer;
* a history of blood clots in the legs or lungs;
* undiagnosed vaginal bleeding;
* porphyria;
* diabetes mellitus;
* malignant melanoma;
* gallbladder or pancreatic disease;
* heart or kidney disease;
* cerebrovascular disease (stroke);
* cigarette smoking;
* a history of suicide attempts or psychotic episodes requiring hospitalization;
* recurrent migraine headaches;
* pregnancy (patients will be warned not to become pregnant during the study and will be required to agree to employ barrier contraceptive methods);
* pregnancy-related medical conditions such as hyperemesis, pre-toxemia and toxemia, deep vein thrombosis (DVT) and bleeding diathesis;

Any woman with a first degree relative (immediate family) with either ovarian cancer, premenopausal breast cancer or breast cancer presenting in both breasts or any woman who has multiple family members (greater than three relatives) with postmenopausal breast cancer will also be excluded from participating in this protocol;

Any woman meeting the Stages of Reproductive Aging Workshop Criteria (STRAW) for perimenopause will be excluded from participation. Specifically, we will exclude any woman with an elevated plasma follicle stimulating hormone (FSH) level (> 14 IU/L) and with menstrual cycle variability of > 7 days different from their normal cycle length.

Ages: 22 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2016-10-13 (Actual); Study Completion 2016-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal E Schiller, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill; David R Rubinow, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloch M, Schmidt PJ, Danaceau M, Murphy J, Nieman L, Rubinow DR. Effects of gonadal steroids in women with a history of postpartum depression. Am J Psychiatry. 2000 Jun;157(6):924-30. doi: 10.1176/appi.ajp.157.6.924. PMID 10831472
- [Derived] Rudzinskas SA, Mazzu MA, Schiller CE, Meltzer-Brody S, Rubinow DR, Schmidt PJ, Goldman D. Divergent Transcriptomic Effects of Allopregnanolone in Postpartum Depression. Genes (Basel). 2023 Jun 8;14(6):1234. doi: 10.3390/genes14061234. PMID 37372414
- [Derived] Rudzinskas SA, Goff AC, Mazzu MA, Schiller CE, Meltzer-Brody S, Rubinow DR, Schmidt PJ, Goldman D. Intrinsically dysregulated cellular stress signaling genes and gene networks in postpartum depression. Mol Psychiatry. 2023 Jul;28(7):3023-3032. doi: 10.1038/s41380-023-01985-5. Epub 2023 Feb 13. PMID 36782063
- See also: University of North Carolina Center for Women's Mood Disorders — http://www.med.unc.edu/psych/wmd

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 3,341 completed screening forms, 406 women appeared initially eligible. 54 were responsive, interested in participating, and eligible to enroll based on pre-screening (unmedicated, without current psychiatric illness or chronic health conditions).
Pre-assignment Details: Of the 54 women who were recruited to participate, 18 did not meet our eligibility criteria during the extensive safety screening phase because of medical conditions found upon exam, use of medications, family history of reproductive cancer, history of pregnancy-related medical condition, and lack of compliance with the screening protocol.
Groups:
- Women With Postpartum Depression (PPD): 4 monthly intramuscular (IM) injections of leuprolide acetate (Lupron) 3.75 mg; micronized estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day; progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day. Participants will also receive placebo.
  Leuprolide Acetate: All subjects will receive one IM injection (3.75 mg) each month for four months.
  Micronized estradiol: All participants will receive micronized estradiol daily for eight weeks. Estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day.
  Progesterone: All subjects will receive micronized progesterone daily for eight weeks. Progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day.
- Women Without Any Psychiatric History (Control): 4 monthly IM injections of leuprolide acetate (Lupron) 3.75 mg; micronized estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day; progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day. Participants will also receive placebo.
  Leuprolide Acetate: All subjects will receive one IM injection (3.75 mg) each month for four months.
  Micronized estradiol: All participants will receive micronized estradiol daily for eight weeks. Estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day.
  Progesterone: All subjects will receive micronized progesterone daily for eight weeks. Progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day.
Period: Overall Study
Arm/Group | Women With Postpartum Depression (PPD) | Women Without Any Psychiatric History (Control)
Started | 19 | 17
Hypogonadism | 18 | 15
Addback | 16 | 15
Withdrawal | 15 | 15
Completed | 15 | 15
Not Completed | 4 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Women With Postpartum Depression (PPD); Women Without Any Psychiatric History (Control): 4 monthly IM injections of leuprolide acetate (Lupron) 3.75 mg; micronized estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day; progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day. Participants will also receive placebo.
  Leuprolide Acetate: All subjects will receive one IM injection (3.75 mg) each month for four months.
  Micronized estradiol: All participants will receive micronized estradiol daily for eight weeks. Estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day.
  Progesterone: All subjects will receive micronized progesterone daily for eight weeks. Progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day.
- Total: Total of all reporting groups
Arm/Group | Women With Postpartum Depression (PPD) | Women Without Any Psychiatric History (Control) | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 17 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.053 (4.916) | 36.294 (4.224) | 35.639 (4.580)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 14 | 11 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Blood-oxygen-level-dependent (BOLD) Response During Functional Magnetic Resonance Imaging (fMRI) z Statistic
Description: The primary outcome measure was functional magnetic resonance imaging (fMRI) data collected during a Monetary Incentive Delay (MID) Task. The BOLD response was examined within the nucleus accumbens, a brain region that responds to monetary rewards. The z statistic represents the maximum contrast between win versus non-win outcomes during the MID task in the nucleus accumbens, averaged across the participants in each group. The mean BOLD response ranged from z=1.7 to 2.3; higher z scores indicate greater activation of the nucleus accumbens during reward. Individual z scores were generated using the Oxford Centre for Functional Magnetic Resonance Imaging of the Brain (FMRIB) software library (FSL), which is a library of brain imaging analysis tools for fMRI.
Time Frame: baseline and hormone withdrawal
Population: Of the 36 women who enrolled in the study, 6 were withdrawn prior to the second fMRI session. For the purpose of this group x time analysis, their data have been excluded. In addition, one participant had significant motion artifact (>4mm) during one run of the MID, and as such, her data were excluded from the analyses.
Measure: Mean (Standard Deviation); unit: z score
Groups:
- Women With a History of Postpartum Depression (PPD); Women Without Any Psychiatric History (Control): 4 monthly IM injections of leuprolide acetate (Lupron) 3.75 mg; micronized estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day; progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day. Participants will also receive placebo.
  Leuprolide Acetate: All subjects will receive one IM injection (3.75 mg) each month for four months.
  Micronized estradiol: All participants will receive micronized estradiol daily for eight weeks. Estradiol will be started at a dose of 4 mg/day and increased progressively up to 10 mg/day.
  Progesterone: All subjects will receive micronized progesterone daily for eight weeks. Progesterone will be started at 400 mg/day and increased progressively up to 800 mg/day.
Arm/Group | Women With a History of Postpartum Depression (PPD) | Women Without Any Psychiatric History (Control)
Number analyzed (Participants) | 14 | 15
z score
  Left Nucleus Acc Baseline | 2.3 (1.13) | 2.0 (.99)
  Left Nucleus Acc Withdrawal | 2.1 (1.20) | 1.7 (.69)
  Right Nucleus Acc Baseline | 2.2 (1.12) | 2.0 (1.09)
  Right Nucleus Acc Withdrawal | 2.3 (1.05) | 2.0 (.83)
Statistical Analysis 1: Comparison: Women With a History of Postpartum Depression (PPD) vs Women Without Any Psychiatric History (Control); Test type: Superiority; p = .27, repeated measures ANOVA; F=1.40, df=2,26

2. Secondary Outcome: Change in Inventory of Depression and Anxiety Symptoms (IDAS) Dysphoria Score
Description: The IDAS Dysphoria Scale consists of 10 items and uses a 5-point Likert-type scale, ranging from 1 to 5 with 1 indicating "not at all" and 5 indicating "extremely". As such, the range of possible scores is 10 to 50. The Dysphoria scale includes items assessing feelings of depression, inadequacy, psychomotor agitation, guilt, discouragement, anhedonia, poor concentration, difficulty with decision-making, psychomotor retardation, and worry. Higher scores indicate greater dysphoria.
Time Frame: Assessed at baseline and post-treatment
Population: Of the 36 women who enrolled in the study, 6 (4 PPD, 2 controls) were withdrawn prior to the second fMRI session. For the purpose of this group x time analysis, their data have been excluded. All 30 subjects who completed the protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Women With a History of Postpartum Depression (PPD) | Women Without Any Psychiatric History (Control)
Number analyzed (Participants) | 15 | 15
units on a scale
  IDAS Dysphoria Baseline | 11.4 (2.20) | 12.7 (3.08)
  IDAS Dysphoria Withdrawal | 15.7 (8.29) | 11.1 (1.34)
Statistical Analysis 1: Comparison: Women With a History of Postpartum Depression (PPD) vs Women Without Any Psychiatric History (Control); Test type: Superiority; p = .018, repeated measures ANOVA; F=6.29, df=1,28

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for every participant over the course of the 7-month-long protocol.
Description: Participants were asked about side effects at every study visit.
Arm/Group | Women With Postpartum Depression (PPD) | Women Without Any Psychiatric History (Control)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 12/19 | 11/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Women With Postpartum Depression (PPD) (N=19) | Women Without Any Psychiatric History (Control) (N=17)
Fatigue (General disorders) | 6 | 6
Spotting/abnormal menstrual bleeding (Reproductive system and breast disorders) | 5 | 2
Nausea and/or vomiting (Gastrointestinal disorders) | 2 | 1
Dizziness (Nervous system disorders) | 5 | 5
Cracked nipple(s) (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hair loss (Skin and subcutaneous tissue disorders) | 1 | 0
Vaginal itching (Reproductive system and breast disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Bradycardia or Arrhythmia (Cardiac disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest pain (Cardiac disorders) | 2 | 0
Difficulty concentrating/memory impairment (Psychiatric disorders) | 0 | 2
Hot flashes (Reproductive system and breast disorders) | 0 | 2
Heartburn or reflux (Gastrointestinal disorders) | 0 | 1
Cramps (Reproductive system and breast disorders) | 0 | 1
Weight gain (General disorders) | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes